CLINICAL TRIAL: NCT03871608
Title: Validation of a Standardized Tool for Evaluation Function of Patients With Temporomandibular Disturbances (DTM) by Physiotherapists
Brief Title: Validation of a Standardized Tool for Evaluation Function of Patients With TMD
Acronym: DTM-SCORE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9865
Record Dates: First submitted 2019-01-08; First posted 2019-03-12 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Temporomandibular Joint Disorders
Keywords: temporomandibular joint disorders; rehabilitation; assessment
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DTM Disorders: Patient with DTM Disorders with Examination of functional etiologies on DTM Disorders and Assessment of symptoms on DTM Disorders
  Interventions: Other: Examination of functional etiologies on DTM Disorders; Other: Assessment of symptoms on DTM Disorders

INTERVENTIONS:
Other: Examination of functional etiologies on DTM Disorders — Evaluating functional etiologies accessible to rehabilitation, consists of 4 categories (Orofacial dyspraxia, parafunctions, posture, Chewing) and includes 11 items in total
Other: Assessment of symptoms on DTM Disorders — Examining the symptoms of the patient, consists of 5 categories (Muscle examination, Areas of cellulalgic infiltrates, Mandibular kinetics, Joint sounds, Thrust)and includes 21 items

SUMMARY:
Temporo-Mandibular Disorders (TMD) are the reason for consultation on more common in maxillofacial. However, there is no consensus on their care. For a long time, Rehabilitative management of the TMD was content to treat only the symptoms.

No validated score does not allow to evaluate globally the malfunctions at the origin of the TDM, as well as the symptoms and functional discomfort that result. The creation of such a tool would standardize the physical examination of the physiotherapist.

This is a functional evaluation scale including 2 subparts: an examination of functional etiologies and an assessment of symptoms. At the same time, a self-questionnaire was created to gather the patient's feelings and evaluate the impact of the TMD on his life daily.

The outcome of this research would be to create a score to track the patient's progress during the reeducation, trying to rate the different factors according to their number and severity. This tool would then make it possible to objectify the impact of rehabilitation treatment on the factors etiological and verify the effectiveness of rehabilitation protocols.

DETAILED DESCRIPTION:
Temporo-Mandibular Disorders (TMD) are the reason for consultation on more common in maxillofacial. However, there is no consensus on their care. For a long time, Rehabilitative management of the TMD was content to treat only the symptoms.

No validated score does not allow to evaluate globally the malfunctions at the origin of the TMD, as well as the symptoms and functional discomfort that result. The creation of such a tool would standardize the physical examination of the physiotherapist.

This is a functional evaluation scale including 2 subparts: an examination of functional etiologies and an assessment of symptoms. At the same time, a self-questionnaire was created to gather the patient's feelings and evaluate the impact of the TMD on his life daily.

The outcome of this research would be to create a score to track the patient's progress during the reeducation, trying to rate the different factors according to their number and severity. This tool would then make it possible to objectify the impact of rehabilitation treatment on the factors etiological and verify the effectiveness of rehabilitation protocols.

Existing tools:

Imaging: If MRI has long been used to verify the effectiveness of management, the emphasisthe weak link between MRI results and functional disorders, dethroned this examination for the benefit of clinical examination.

Currently, several scores are validated :

- Helkimo Index = Craniomandibular Dysfunction Index (CDI): Objectives: This is an epidemiological index, developed in 1974 by Helkimo, to assess the needs of treatment in the population by measuring the severity of the symptoms. It provides a good indication of the severity of the TMD. It is still used today in studies.

Limitations of use: It was not designed to evaluate the effectiveness of a rehabilitative management. This diagnostic test of the TMD makes it possible to classify the patients according to the severity of the symptoms but provides no indication of etiological

- Craniomandibular Index (CMI): Objectives: This index was created in 1985 by Fricton and Schiffman for use in both studies epidemiological and clinical. It measures the variations of the TMD and can therefore be used in the studies evaluating therapeutic strategies [10]. It is divided into two parts: the DI (dysfunction index) and the PI (Palpation index). Limitations of use: However, following the evolution of the management of the TMD, the CMI score presentssome limits. Indeed, this index lists and evaluates the different symptoms of the patient sodetailed (mandibular kinetics, joint sounds and muscle palpation). But, this score does not take into account the new etiologies, it does not make it possible to evaluate the impact of their rehabilitative treatment on the result.

- DRC / TMD (Research Diagnostic Criteria for Temporomandibular Disorders): Objectives: In 1992, Dworkin et al. have established diagnostic criteria for research for disorders temporomandibular devices (DRC / TMD) to provide a reliable diagnostic tool. The goal was to develop a set of diagnostic criteria for TMD. It includes 2 axes: an interrogation and a physical examination. This score was translated into French in 2002. This is the only existing score taking into account the impact of TMD on the patient's life (functional impairment in daily life).

Limitations of use: Although it evaluates certain etiologies (psychological factors and bruxism), it neglects however all functional etiologies. Moreover, being very detailed, its implementation is time-consuming and makes it difficult to use in everyday practice.

Psychometric benefits and limitations:

Metric values showed acceptable high reliability (except for diduction). The reliability of the extra-oral palpation is correct or elevated. However, the inter-examiner reliability of the Intraoral palpation is weak. This is partly because the examination includes palpation of the Lateral pterygoid, but this one is inaccessible to palpation according to several studies.

- Palpation test (Palp-Test): Objectives: This is a palpation index of 20 sites involved in the TMD. The test has the advantage of being fast and only takes a minute to complete.

Limitations of use: The disadvantage of this score is that it is restricted. It does not reflect the totality of the symptomatology of the patient.

This assessment tool presented in the form of a functional review and a self-questionnaire fill the gaps presented in existing scores, by bringing new prospects. In addition to assessing the symptoms of the patient, this tool created takes into account etiologies responsible for the appearance and maintenance of the pathology. The self-questionnaire, to be completed by the patient, allows you to evaluate your feelings in order to highlight the impact of TMD on your daily life.

ELIGIBILITY:
Specific Inclusion criteria :

* Patients consulting for DTM at the CHU of Montpellier within the CMF service
* Results obtained with the Helkimo score: moderate to severe
* Age range: between 18 and 75 years old included

Non-specific inclusion criteria:

* Collection of informed written consent of the patient
* Affiliation or beneficiary of a social security scheme

Non-specific exclusion criteria:

* Patient under tutorship or curatorship
* Patient under the protection of justice

Specific exclusion criteria:

* Not included for assessment difficulty:

  * Associated disease or disability that can skew assessments
  * Diseases causing neurological (facial paralysis) or rheumatic (Spondyloarthritis) ankylosing, rheumatoid arthritis) with consequence on TMJ temporomandibular disturbances appeared following a trauma
  * Failure to understand questions or instructions
* No inclusion for no indication of rehabilitation:

  * Large facial dysmorphoses (ODF treatment or surgery)
  * Loss of posterior wedging uncompensated (restoration in odontology)
* Exclusion for tracking difficulties:

  * Lack of motivation of the patient
  * Mutation or planned move

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with TMD Disorders
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Validation of the assessment tool | 40 months
  Validate an assessment tool for diagnosis of functional etiologies including oroficial dyspraxia, respiration dyspraxia (oral or combined), labial dyspraxia and lingual dyspraxia (lingual immaturity and swallowing dysfunction)
Establishment of a symptom score | 40 months
  Validate an assessment tool to score the evolution of the patient with DTM. It's to evaluate the crackles of the jaw, the pain and the dyskinesia.

SECONDARY OUTCOMES:
Evaluation of the acceptability of the assessment tool | 40 months
  The rate of unfilled items will be described, The ceiling and floor effects, The filling time of the 2 parts of the questionnaire, Study of the redundancy between items by the correlation between items
Evaluation of the Reproducibility inter-observer of the assessment tool | 40 months
  Evaluating the initial balance sheet will be compared between the 2 independent physiotherapists. The concordance of these 2 assessments will be estimated in order to measure inter-observer reproducibility.
Evaluation of the Reproducibility intra-observer of the assessment tool | 40 months
  Compare the 2 assessments of the same physiotherapist at the initial assessment and 7 days after (just before the rehabilitation).
Internal validity of the scale of the assessment tool | 40 months
  Assess whether changes in the results obtained with the assessment tool about the evaluation of the symptoms are a real change or are related to the evaluator (intra-examiner assessment)
External validity of the assessment tool | 40 months
  Evaluation of the correlation (items and scores) between the assessment tool and the Scale Research Diagnostic Criteria for Temporomandibular Disorders (RDC / TMD) and evaluating the discriminant validity, ability of the scale to distinguish different grades of severity from TMD or different levels of pain and discomfort
Sensitivity to change of the assessment tool | 40 months
  Evaluation of the pain by the EVA scale mesured at the initial and final visit and comparison with the symptomatology part of the assessment tool
Sensitivity to change of the assessment tool | 40 months
  Evaluation of the functional impairment by the EVA scale mesured at the initial and final visit and comparison with the symptomatology part of the assessment tool
Sensitivity to change of the assessment tool | 40 months
  Evaluation of the quality of life by the EVA scale mesured at the initial and final visit and comparison with the symptomatology part of the assessment tool

CONTACTS AND LOCATIONS:
Overall Officials: Patrick JAMMET, PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Hôpital Gui de Chauliac, Montpellier, France

IPD SHARING:
Plan to Share IPD: No